CLINICAL TRIAL: NCT05232994
Title: Use of Combination Metformin and Esomeprazole in Preterm Pre- Eclampsia: Randomized Controlled Trial
Brief Title: Metformin and Esomeprazole For Preterm Pre-eclampsia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DDD# 605095
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Preeclampsia Severe; Preeclampsia Second Trimester; Preterm Birth Complication
MeSH Terms: interventions — Esomeprazole; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- combination metformin and esomeprazole (Experimental): Combination 2 g of oral extended release metformin, in divided doses and Esomeprazole 20mg daily until delivery.
  Interventions: Drug: Esomeprazole 20mg
- expectant management (No Intervention)

INTERVENTIONS:
Drug: Esomeprazole 20mg — Combination 2 g of oral extended release metformin, Esomeprazole 20mg daily until delivery.
  Other Names: Metformin
  Arms: combination metformin and esomeprazole

SUMMARY:
A recent randomized controlled trial by Cluver et al included 180 women with preterm pre-eclampsia between 26+0 to 31+6 weeks' gestation undergoing expectant management: 90 were randomised to extended release metformin and 90 to placebo. Investigators found that extended release metformin (3g daily) can prolong gestation in women with preterm pre-eclampsia. Combination metformin and esomeprazole has shown promise in the treatment of preeclampsia as both agents reduce placental and endothelial secretion of soluble fms-like tyrosine kinase 1 (sFlt-1) and soluble endoglin, and reduce endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Individuals presenting with pre-eclampsia between 24+0 and 31+6 weeks of gestation, with a single viable fetus and no major anomalies

* Women 18 years or older
* Women diagnosed with preeclampsia
* Women with pre-eclampsia superimposed on chronic hypertension
* Candidates for expectant management and had no clinical indication for immediate delivery

Exclusion Criteria:

* Delivery within 48hr is highly likely
* Maternal or fetal compromise that necessitated immediate delivery
* Diabetes or gestational diabetes currently on metformin therapy
* Contraindications to metformin, esomeprazole
* Baseline creatinine >124 μmol/L
* Hypersensitivity to metformin or esomeprazole
* Metabolic acidosis
* Use of drugs that might interact with metformin (glyburide, furosemide, or cationic drugs) Multiple gestations

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mean plasma difference in sFlt-1 from randomization to day 7 | from randomization to day 7

SECONDARY OUTCOMES:
Mean plasma difference in vascular endothelial growth factor (VEGF) | from randomization to day 7
Mean plasma difference in placental growth factor (PlGF) levels | from randomization to day 7
Mean plasma difference in soluble endoglin (sEng) | from randomization to day 7
Maternal death | At time of delivery
Mean highest blood pressure during expectant management mmHg | At time of delivery
Number of anti-hypertensive medications at delivery | at time of delivery
Fetal growth restriction defined as a sonographic estimated fetal weight (EFW) or abdominal circumference (AC) below the 10th percentile for gestational age using Hadlock cutoffs | at time of delivery
Gestational age at delivery | at time of delivery
Neonatal intensive care unit (nicu) admission | at time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hoffman, MD, MPH, Principal Investigator — ChristianaCare
Locations (1):
- Christiana Care Health Systems, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data are available for 5 years at a third party website